



# **GOLD AF**

Registry

# Statistical Analysis Plan

Version 1.1

19.12.2018

Sponsor: Medtronic International Trading Sàrl, Route du Molliau 31 CH-1131 Tolochenaz Switzerland

CRO:
IHF GmbH - Institut für Herzinfarktforschung
Bremserstraße 79
67063 Ludwigshafen/Rhine
Germany

# **Signature Page**

We, the undersigned, have carefully read this Statistical Analysis Plan and agree that it contains all necessary information required for statistical analyses of the GOLD AF registry:

| Signature | Date |
|---|---|
| Ocm &A Ekaterina Ostern Clinical Study Manager Medtronic International Trading Sàrl | 18, Jan, 2019 |
| Juliane Karthe Project Manager IHF GmbH - Institut für Herzinfarktforschung | M. JAN2013 |
| Tobias Müller EBogen Programmer / Data Management Responsible IHF GmbH - Institut für Herzinfarktforschung | 02.JAN 2019 |
| Martin Horack | 12 DECEOIS |

Biostatistician

IHF GmbH - Institut für Herzinfarktforschung

# **Version History**

| Version | Date | Author | Changes |
|---|---|---|---|
| DRAFT<br>Versions | 13.05.2015 | Dr. Alexandra Bernhardt<br>Martin Horack | Initial development |
| Version<br>1.0 | 31.08.2017 | Martin Horack | Update, minor changes |
| Version<br>1.1 | 21.12.2018 | Christiane Lober<br>Martin Horack | definition changes in Analysis sets, adapt to updated FU windows and handling follow-ups, add analysis specifications and details in endpoint relevant calculations, add subgroup analysis and comparisons (appendix), adding EFAS (analysis set) Updates according to Quality Meeting of 25th of October 2018 |

# **Table of Contents**

| Signatu | re Page | | 2 |
|---|---|---|---|
| Version | History | | 3 |
| Table of | Contents | | 4 |
| Abbrevi | ations | | 6 |
| 1<br>1.1<br>1.2<br>1.3 | General Infor<br>Statistical Site | mation | 9<br>10 |
| 2<br>2.1<br>2.2 | Main Objectiv | the Non-interventional Study<br>/e<br>pjectives | 11 |
| 3<br>3.1<br>3.2<br>3.3 | Design<br>Flow Chart | Determination | 12<br>13 |
| 4<br>4.1<br>4.2<br>4.3<br>4.4 | All-Documen<br>Baseline Anal<br>Full Analysis S | ted Patient Set<br>ysis Set<br>Set<br>Analysis Set | 16<br>16<br>16 |
| 5 | , . | he EFAS will be used in the same way as the FAS.Protocol | 18 |
| 6<br>6.1<br>6.2<br>6.3<br>6.3.1 | Study Popula<br>Analysis Varia<br>Quality of Life | lestionbles | 19<br>19<br>19 |
| 7<br>7.1<br>7.2<br>7.2.1<br>7.2.2<br>7.2.3<br>7.2.4<br>7.3<br>7.4<br>7.4.1<br>7.4.2<br>7.4.3<br>7.5 | Definitions Handling data Patient data Procedural da Follow-up da Adverse Even Categorisatio Transformatic (Re-)Calculati Risk scores Scoring of qu | ga entity types | |
| 7.5.1 | | of missing values | |

| 7.5.2 | Replacement of outliers | 32 |
|---|---|---|
| 7.6 | Self-Evident Corrections | |
| 8 | Descriptive Statistics | 33 |
| 8.1 | Statistical analyses for the main objective | 34 |
| 8.1.1 | Estimate Phased RFA 12 month success rate | 34 |
| 8.1.2 | Methodology for analysing the main objective | 36 |
| 8.2 | Statistical analyses for additional objective | 37 |
| 8.2.1 | Estimate Phased RFA procedure safety | |
| 8.2.2 | Methodology for analysing the procedure safety | 39 |
| 8.3 | Statistical analyses for ancillary objectives | |
| 8.3.1 | Characterize the acute procedural success rate | |
| 8.3.2 | Assess Phased RFA efficiency | |
| 8.3.3 | Characterize the peri-procedural anticoagulation therapy | |
| 8.3.4 | Describe single catheter PVAC GOLD utilization in persistent AF | |
| 8.3.5 | Evaluate QoL (AFEQT) dynamic at 12 month FU | |
| 8.4 | Interim analysis | |
| 8.5 | Final analysis | |
| 8.6 | Analysis of group comparisons and subgroups | |
| 8.6.1 | Analysis of subgroups | |
| 8.6.2 | Analysis of comparison groups | |
| 8.7 | Benchmark reports | |
| 8.8 | Graphical analysis | 45 |
| 9 | References | 47 |
| Append | dix A: Table specifications (examples) | 48 |
| Append | dix B: Analysis tables, Study objectives and Analysis sets | 49 |
| Append | dix C: Subgroup analysis | 51 |
| Append | dix D: Analysis of comparison groups | 53 |
| Append | dix E: Annotated eCRF V1.3 and V1.4 | 55 |
| Annend | dix F. Follow-up Re-Assignment | 56 |

# **Abbreviations**

| 12MFU | 12 months follow-up |
|---|---|
| ACE inhibitors | Angiotensin-Converting |
| ACT | Activated Clotting Time |
| AE | Adverse Event |
| AF | Atrial Fibrillation |
| AFEQT | Atrial Fibrillation Effect on Quality of Life (Questionnaire) |
| Afl | Atrial Flutter |
| ASA | AcetylSalicylic Acid |
| AT II antagonist | Angiotensin Receptor II Antagonist |
| AV-Block | AtrioVentricular Block |
| CABG | Coronary Artery Bypass Graft |
| CFAE | Complex Fractionated Atrial Electrograms |
| cGy | CentiGray |
| CHA2DS2-VASc | Score for Stroke Risk |
| CHAZD3Z-VA3C | Components: cardiac failure,hypertension, age ≥75 (doubled), diabetes, stroke (doubled)-vascular disease, age 65–74 and sex category (female) |
| CI | Confidence Interval |
| CIP | Clinical Investigational Plan |
| cm | Centimeter |
| COPD | Chronic Obstructive Pulmonary Disease |
| CRF | Case Report Form |
| CRO | Contract Research Organisation |
| CRT | Cardiac Resynchronization Therapy |
| CT | Computed Tomography |
| CV | Cardio Version |
| CVD | Cardiovascular Disease |
| DAP | Dose Area Product |
| dd.mm.yyyy | Date with Day.Months.Year |
| EBogen | Electronic Data Capture System of the Institut für Herzinfarktforschung |
| ECG | Electrocardiogram |
| eCRF | Electronic Case Report Form |
| EDC | Electronic Data Capture |
| EGM | Electrogram |
| EHRA | European Heart Rhythm Association |
| EP | Electrophysiology |
| FU/GFU | Follow-up/General Follow-up |
| GmbH | Gesellschaft mit beschränkter Haftung (limited liability company) |
| HAS-BLED | Score for Major Bleeding Risk |
| | Components: hypertension, abnormal renal/liver function (1point each), stroke, bleeding history or predisposition, labile INR, elderly (>65), Drugs/alcohol concomitantly (1 point each) |
| HF | Heart Failure |
| hh:mm | Time with Hours.Minutes |
| ICD | Implantable Cardioverter-Defibrillator |
| ICM | Implantable Cardio Monitor |
| IHF | IHF GmbH - Institut für Herzinfarktforschung, Ludwigshafen |

| ILR | Implantable Loop Recorder |
|---------------------|--------------------------------------|
| INR | International Normalized Ratio |
| IPG | Implantable Pulse Generator |
| IVC | Inferior Vena Cava |
| kg | Kilogram |
| LA | Left Atrium |
| LAAO | Left Atrial Appendage Occluder |
| LCPV | Left Common Pulmonary Vein |
| LIPV | Left Inferior Pulmonary Vein |
| LMWH | Low-Molecular-Weight Heparin |
| LSPV | Left Superior Pulmonary Vein |
| LV | Left Ventricle |
| LVEF | Left Ventricular Ejection Fraction |
| MAAC | Multi-Array Ablation Catheter |
| MASC | Multi-Array Septal Catheter |
| MDT | Medtronic |
| mGy*cm <sup>2</sup> | MilliGray Square Centimeters |
| MI | Myocardial Infarction |
| min | Minute |
| ml | Milliliter |
| mm | Millimeters |
| mmHg | Millimeters of Mercury |
| MRI | Magnet Resonance Imaging |
| NA | Not Applicable |
| NIS | Non-interventional Study |
| no. | Number |
| NOAC | Novel Oral Anticoagulant |
| NSAID | NonSteroidal Anti-Inflammatory Drugs |
| NSR | Normal Sinus Rhythm |
| NYHA | New York Heart Association |
| Ор | Operator |
| PAF | Paroxysmal Atrial Fibrillation |
| PCI | Percutaneous Coronary Intervention |
| PDRF | Patient Data Release Form |
| PIC | Patient Informed Consent |
| PV | Pulmonary Vein |
| PVAC | Pulmonary Vein Ablation Catheter |
| PVI | Pulmonary Vein Isolation |
| Q1 | Lower Quartile |
| Q3 | Upper Quartile |
| QoL | Quality of Life |
| RA | Right Atrium |
| RF | Radiofrequency |
| RFA | Radiofrequency Ablation |
| RIPV | Right Inferior Pulmonary Vein |
| RMPV | Right Middle Pulmonary Vein |
| RSPV | Right Superior Pulmonary Vein |
| SAE | Serious Adverse Event |

| SAP | Statistical Analysis Plan |
|-----|-----------------------------------|
| SAS | Statistical Analysis System |
| SD | Standard Deviation |
| sec | Second |
| SVC | Superior Vena Cava |
| TEE | Trans-Esophageal Echocardiography |
| TIA | Trans-Ischaemic Attack |
| TTE | Trans-Thoracic Echocardiogram |
| VF | Ventricular Fibrillation |
| VKA | Vitamin K Antagonist |
| VT | Ventricular Tachycardia |

# 1 Introduction

#### 1.1 General Information

The intention of this Statistical Analysis Plan is to specify procedures regarding all planned statistical analyses within the framework of the GOLD AF registry performed by the IHF GmbH - Institut für Herzinfarktforschung, Ludwigshafen. The overall objective of the SAP is to ensure the credibility of the study data by describing the statistical methodology to be used to evaluate the baseline and follow-up data of the GOLD AF registry.

The initial version of the Statistical Analysis Plan will be completed before first database lock. However, any of the following points may become subject to alterations during the course of the study. Significant changes to statistical analyses shall be discussed with the Statistical Analysis Plan approvers prior to their implementation. All parties affected by changes are to be informed by the author of the changes.

If necessary, selected tasks may be delegated to authorised and adequately qualified designees by the assigned personnel without the need to update the Statistical Analysis Plan. However, the responsibilities remain with the personnel assigned in the Statistical Analysis Plan.

By the time of database lock, the Sponsor Project Responsible shall receive the final version of the Statistical Analysis Plan.

This is a non-interventional registry. The statistical analysis will be performed on an exploratory and descriptive basis and there are no initial hypotheses to be tested.

This Statistical Analysis Plan has been written based on the following documents for this prospective non-interventional registry GOLD AF:

- o Clinical Investigational Plan (Version 1.0 dated 06-Feb-2015)
- o Clinical Investigational Plan (Version 2.0 dated 09-Sept-2016)
- o Case Report Form (Version 1.3 dated 30-APR-2015)
- o Case Report Form (Version 1.4 dated 13-Jan-2017)
- Annotated Case Report Form (Version 1.3) Appendix E
- Annotated Case Report Form (Version 1.4) Appendix E
- o Data Management Plan (V1.2 dated 05-Jul-2016)
- o Online Data Validation Plan (V1.0 dated 21-SEP-2015)

## 1.2 Statistical Site

The statistical analysis of this registry will be performed by the following Contract Research Organisation (CRO):

#### IHF GmbH – Institut für Herzinfarktforschung

Bremserstr. 79, 67063 Ludwigshafen/Rhine, Germany Phone: +49 621 59577 222 FAX: +49 621 59577 400

The responsible CRO statistician is:

Martin Horack Phone: +49 621 59577 210 FAX: +49 621 59577 410 Email: horack@ihf.de

## 1.3 Software

Statistical analysis will be carried out using SAS®, release 9.3 or higher (SAS Institute Inc., Cary, NC, USA) on a Microsoft® Windows® 7 or a Microsoft® Windows® 10 Enterprise platform.

# 2 Objectives of the Non-interventional Study

## 2.1 Main Objective

The primary objective of this study is to assess the Phased RF ablation success rate after 12 month follow-up in patients with AF who are scheduled for Phased RFA.

# 2.2 Secondary Objectives

Ancillary objectives of this study are as follows:

- Estimate Phased RFA safety
- Characterize the acute procedural success rate
- Assess Phased RFA efficiency
- Characterize the peri-procedural anticoagulation therapy
- Describe single catheter PVAC GOLD utilization in persistent AF
- Evaluate QoL ("AFEQT" questionnaire)

# 3 Study Design

# 3.1 Design

The GOLD RF registry is a postmarket release (PMR), prospective, observational, multicentre, clinical study in consecutive subjects with atrial fibrillation treated with the phased RFA technology (Medtronic, Minneapolis, MN, USA). Patient's participation in this study has no impact on his or her indication, diagnostics or therapy. Subjects are supposed to be treated in compliance with current valid Instructions for Use (IFU) as well as according to medical society guidelines and the clinic's internal directives. Medication-based therapy should also meet medical society guidelines or the clinic's internal directives, respectively.

40 sites in 14 countries (Germany, Netherlands, United Kingdom, Hungary, Italy, Spain, Switzerland, Israel, Poland, Portugal, France, Greece, Georgia and South Korea) are anticipated to take part in the registry to get documentation on at least 800-1000 patients (for more details regarding sample size consideration, see Section 3.3 in the SAP). Eligible for participation are study sites and hospital-based physicians treating AF subjects with phased RFA technology. The enrolment period is estimated to be 24 months. The individual observation period per patient is up to 12 (+2) months: Based on the observational plan, it is planned that the baseline visit is conducted by the investigators. All follow-up visits in the registry are unscheduled. They will be conducted in accordance with "routine clinical practice" in the participating medical centres: Between the procedure date and the following 12MFU period, any general FU will be captured. General FUs might occur due to site specific visit schedule, related to AF re-occurrence (re-ablation, AF symptoms, CV etc.) or due to patient visits at the site because of AE related symptoms. At 12MFU window, the patient will either be followed up in the medical centre or by phone.

# 3.2 Flow Chart

| | | Procedure | Canaval | 12 months | 12 months |
|---|---|---|---|---|---|
| Data Collection* | Baseline | first docu-<br>mented,<br>additional | General<br>Visit/ FU | FU<br>in hospital | FU<br>by phone |
| Enrolment (PIC/PDRF) | Χ | | | | |
| Demographics | X | | | | |
| Medical History <sup>#</sup> | X | | | | |
| Concomitant disease | X | | | | |
| Diagnostics | X | | X | X | Х |
| Symptoms | | | X | X | X |
| Medication list | X | | × | X | X |
| Administrative information | | X | X | X | Х |
| Anticoagulation pre-intra-<br>procedural | | X | | | |
| General procedure summary | | X | | | |
| Consumables | | X | | | |
| PVI confirmation | | X | | | |
| Hospital discharge | | X | | | |
| Quality of Life (AFEQT) | Х | | | X | Х |
| History of AF since last visit | | | X | Х | Х |
| Hospitalization | | | X | X | Х |
| Adverse events (AEs) | - Whenever | occur - | <u> </u> | 1 | |

<sup>\*=</sup> prior to first patient enrolment every site needs to fill in a site questionnaire once

<sup>#=</sup> Medical history includes questions about prior CVD, history of AF, main underlying disease, concomitant disease and history of AF.



Figure 1: Study design – flow chart.

# 3.3 Sample Size Determination

The sample size calculation is based on the main objective to document real life mid-term efficacy of patients with atrial fibrillation who were scheduled for phased RF ablation. Efficacy is in this case assumed as the proportion of redo ablations 12 months after treatment

The table below shows the sample size needed for estimating a binomial proportion for given prevalence with corresponding precision.

 Table 1: Cross table for precision and prevalence for sample size assessment.

| | Precision | | | |
|------------|-----------|------|-----|-----|
| Prevalence | 1% | 2.5% | 5% | 10% |
| 0.1 | 4150 | 665 | 167 | 42 |
| 0.2 | 7377 | 1181 | 296 | 75 |
| 0.3 | 9682 | 1550 | 388 | 98 |

Precision = half-width of a 95% CI

Design effect = 1.2 (variance inflation due to cluster sampling design) Low sampling rate assumed to have no impact on sample size calculation Assuming a prevalence of re-ablation 12 months after treatment of 20%, a sample size of 800 will allow the study to estimate the prevalence with a given precision of  $\pm$  3.8% [range of 95%-CI: 7.6%]. This size guarantees sufficient information to estimate the prevalence in smaller subgroups (e.g. subgroup with a prevalence of 25% with a precision of  $\pm$  6.6% [range of 95%-CI: 13.3%]).

A drop-out rate of 25% is assumed (i.e. an estimated drop-out of about 200 patients). Thus, it is planned to enrol a total number of patients of at least 800 - 1000.

# 4 Analysis Sets

Analysis sets will be predefined and selected for each analysis to be carried out, based on the scope of the analysis. The Appendix B will give an overview about analysis tables, study objectives and analysis sets. Analysis sets might be used for further analysis. The following analysis sets will applied:

## 4.1 All-Documented Patient Set

The All-Documented Patient Set (APS) consists of all patients with signed patient informed consent (PIC) and complete date of PIC who have any additional eCRF documentation, i.e. with non-empty eCRF information for at least one further collection point. In case of a missing PIC/PDRF or an incomplete date of PIC/PDRF, the entry for that patient in the database is only formally created and no further information (at least on further eCRF pages) can be added.

In case that a given PIC/PDRF is drawn back during the course of the registry (i.e. PIC/PDRF is set from "yes" to "no" during the visit), entries that have already been made are not deleted. These entries should be set to missing in the analysis data sets.

If a patient exits from the study, data collected prior to the study withdrawal will be included in the analysis in compliance with PIC/PDRF unless the patient object and ask for deletion of the data or when required by local regulations.

The APS will be used for total registry analysis (interim, final and post-hoc analysis).

# 4.2 Baseline Analysis Set

The Baseline Analysis Set (BAS) consists of all patients of the APS and patients:

- where baseline signature has been taken (signed eCRF)
- with AF who are scheduled for Phased RFA
- that meet all remaining eligibility criteria
- provide any further documentation at baseline
- a phased RFA procedure was started procedure form was fulfilled at least: date of the procedure, PVAC GOLD catheter used (opened), number of PV applications > 0
- patient did not exit the study prematurely for the reason: Patient were enrolled, but
   Phased RFA procedure was not started

According to the Appendix B, the BAS will be used for the interim and final analysis as well as for post-hoc analysis. The final analysis includes the additional objective (SAP chapter 8.2) and ancillary objectives (SAP chapter 8.3), where the BAS will be applied.

# 4.3 Full Analysis Set

The *Full Analysis Set* (FAS) consists of all patients of the BAS and thereof patients with a valid 12MFU form of 12 months visit or 12 months telephone interview. The rules for valid 12MFU form are described in the chapter 7.2.3.

A documented 12MFU form includes at least:

- Date of the visit/FU and
- Vital status and
- Signed eCRF 12MFU visit or 12MFU by phone form

The FAS will be used to analyse the main objective (SAP chapter 8.1), additional objective (SAP chapter 8.2) and ancillary objectives (SAP chapter 8.3). The FAS will be analysed at the end of this study.

# 4.4 Extended Full Analysis Set

The Extended Full Analysis Set (EFAS) consists of all patients of the FAS and thereof patients without documented AF re-ablation (each ablation technology i.e. additional GOLD-AF procedure) until the 12MFU (<351d after the first documented procedure). Also, only patients with a successful first documented procedure (by PVI confirmation) will be member of the EFAS. This population will be used to evaluate the effect of the first documented procedure, in a clearer way.

# 5 For analysis, the EFAS will be used in the same way as the FAS.Protocol Violations

In this registry, the analysis is limited to patients with signed patient informed consent and complete date of patient informed consent (otherwise no further entry in the eCRF was possible) who are scheduled for Phased RFA for AF catheter ablation treatment. Furthermore, the patients have to fulfil the eligibility criteria of an age ≥18 years as well as a signed PIC/PDRF which allows the analysis of collected personal data during the participation in the registry (up to 14 months after the initial Phased RFA procedure). CRF forms documented 14 months after procedure (440 days) will be ignored for analysis.

In this registry it is not distinguished between a broader full analysis set and a more compliant per-protocol set that excludes all major violators. Therefore, the definition of major violators is not applicable.

# **6** Target Variables

## 6.1 Study Population

Data from all patients who are enrolled in the study (patients who meet the eligibility criteria and signed the PIC/PDRF) will be included in the analysis. If a patient exits from the study, data collected prior to the study withdrawal can be included in the analysis in compliance with PIC/PDRF unless patient requests deletion of the personal data when exit the study in compliance with local regulations.

The following parameters will be used to characterise the study population and to give an overview on the documented visits:

- Overview about patient status
  - o number of patients in the All-Documented Patients Set (APS),
  - o number of patients in Baseline Analysis Set (BAS),
  - o number of patients in Full Analysis Set (FAS)
  - o number of patients in Extended Full Analysis Set (EFAS)
- o Overview about reasons for being excluded from the different analysis sets
  - Criteria for the BAS
  - Criteria for the FAS
- Number of documented patients per site (BAS)
- Number of documented patients per visit and visit period (FAS)
- Number of documented visits per patient (FAS)
- o Number of documented patients by visit pattern (FAS)

A patient is defined as "documented" at a respective visit, if the FU form has a date of the visit and it is non-empty (at least one further entry) for that visit.

## 6.2 Analysis Variables

All appropriate information of the following eCRF sections will be used to characterise the study populations (see Appendix D: Annotated Case Report Form V1.3 and V1.4). Data will be displayed based on their entity type (SAP chapter 7.2).

- Demographics and other Baseline Characteristics, Procedure Documentation
- Follow-up Documentation: General FU
- Follow-up Documentation: 12 Months FU
- Follow-up Documentation: 12MFUby Phone
- Adverse Event Form (SUO form)
- Study Exit Form

19.12.2018

Quality of Life Questionnaires

# 6.3 Quality of Life Questionnaires

In this registry, QoL will be assessed with the *Atrial Fibrillation Effect on Quality of Life* (AFEQT) questionnaire. It is a standardized, disease-specific, reliable and responsive measure of health-related QoL in patients with atrial fibrillation. The AFEQT is a self-reported

Institut für Herzinfarktforschung

questionnaire with responses on a 7-point Likert scale. The 20-item instrument is divided into three domains (a 4-item Symptom score, an 8-item Daily Activities score, a 6-item Treatment Concerns score) plus two Treatment Satisfaction questions. The domains Symptoms, Daily Activities and Treatment can be aggregated into an overall score.

For all questionnaires, the frequencies of the given answers are presented by country and overall. If - based on the answers – scores are constructed these are presented, too.

The AFEQT questionnaire consists of 3 functional subscales (Symptoms [4 items], Daily Activities [8 items], Treatment Concern [6 items]) that are part of the overall AFEQT score. The 2 questions on Treatment Satisfaction are computed as its own subscale similarly to the overall score.

- Symptoms [not at all bother OR I did not have this symptom; hardly bothered; a little bothered; moderately bothered; quite a bit bothered; very bothered; extremely bothered]:
  - o Palpitations: Heart fluttering, skipping or racing
  - o Irregular heartbeats
  - Pause in heart activity
  - o Light-headedness or dizziness
- o Daily Activities:
  - Ability to have recreational pastimes, sports, and hobbies
     [not at all limited; hardly limited; a little limited; moderately limited; quite a bit limited; very limited; extremely limited]
  - Ability to have a relationship and do things with friends and family [not at all limited; hardly limited; a little limited; moderately limited; quite a bit limited; very limited; extremely limited]
  - Doing any activity because you felt tired, fatigued, or low on energy [no difficulty at all; hardly any difficulty; a little difficulty; moderately difficulty; quite a bit of difficulty; a lot of difficulty; extreme difficulty]
  - Doing physical activity because of shortness of breath
     [no difficulty at all; hardly any difficulty; a little difficulty; moderately difficulty; quite a bit of difficulty; a lot of difficulty; extreme difficulty]
  - Exercising
     [no difficulty at all; hardly any difficulty; a little difficulty; moderately difficulty; quite a bit of difficulty; a lot of difficulty; extreme difficulty]
  - Walking briskly
     [no difficulty at all; hardly any difficulty; a little difficulty; moderately difficulty; quite a bit of difficulty; a lot of difficulty; extreme difficulty]
  - Walking briskly uphill or carrying groceries or other items, up a flight of stairs without stopping
     [no difficulty at all; hardly any difficulty; a little difficulty; moderately difficulty; quite a bit of difficulty; a lot of difficulty; extreme difficulty]
  - Doing vigorous activities such as lifting or moving heavy furniture, running, or participating in strenuous sports like tennis or racquetball [no difficulty at all; hardly any difficulty; a little difficulty; moderately difficulty; quite a bit of difficulty; a lot of difficulty; extreme difficulty]
- o <u>Treatment Concern</u> [not at all bother; hardly bothered; a little bothered; moderately bothered; quite a bit bothered; very bothered; extremely bothered]:

- o Feeling worried or anxious that your atrial fibrillation can start anytime
- Feeling worried that atrial fibrillation may worsen other medical conditions in the long run
- o Worrying about the treatment side effects from medication
- Worrying about complications or side effects from procedures like catheter ablation, surgery, or pacemaker therapy
- Worrying about side effects of blood thinners such as nosebleeds, bleeding gums when brushing teeth, heavy bleeding from cuts, or bruising
- Worrying or feeling anxious that your treatment interferes with your daily activities
- <u>Treatment Satisfaction</u> [extremely satisfied; very satisfied; somewhat satisfied; mixed with satisfied and dissatisfied; somewhat dissatisfied; very dissatisfied; extremely dissatisfied]:
  - o How well your current treatment controls your atrial fibrillation
  - The extent to which treatment has relieved your symptoms of atrial fibrillation

For the scoring of the AFEQT, see chapter 7.4.3 in the SAP.

#### 6.3.1 Ensure AFEQT data quality for analysis

The following test procedure is planned to admit the use of the AFEQT questionnaire in the GOLD AF registry. Prior analysis, possible effects are needed to discover regarding the following issues:

- a. the use of AFEQT data from not validated language versions
- b. the use of AFEQT data that were not self-administered by the patients, but documented by sites in telephone interviews.

#### Step 1: Validated and not validated AFEQT language versions

The following language versions used in this registry are validated: French, German, Italian, Spanish, Polish, Dutch, English and Korean. The following language versions used in this registry are <u>not</u> validated: Georgian, Greek, Hungarian, Hebrew, Arabic, Russian and Portuguese.

To evaluate whether validated and not validated language versions differ from each other, baseline AFEQT scores will be compared between both groups, i.e. evaluation of homogeneity of both distributions (Wilcoxon-Mann-Whitney test, two tailed, p<0.05). It will be assumed, that both patient sets are equal in their medical history. Further predictors or confounders will not be considered. If the difference proves to be statistically significant, data derived from not validated language versions will be excluded from further analyses. Otherwise, step 2 will be evaluated.

#### Step 2: Self-administered and interview data

The AFEQT was developed and validated as a self-administered questionnaire. However, a currently unknown number of AFEQT questionnaires (i.e. especially those documented during hospital visits) will be collected by the sites and at the 12 months follow-up by phone AFEQT questionnaires will be documented during telephone interviews.

To evaluate whether self-administered and interview data differ from each other, data from both groups (self-administered vs. interview) will be compared (i.e. evaluation of homogeneity of distributions, Wilcoxon-Mann-Whitney test, two tailed, p<0.05). If the difference proves to be statistically significant, data from both groups will not be merged, but analysed separately.

#### Structure and consequences of planned tests:

Scenario 1: Statistically significant difference between validated and not validated language versions

→ Exclusion of data from not validated language version from all further analyses

Scenario 2: No statistically significant difference between validated and not validated language versions

→ Merging and release AFEQT data for step 2

Scenario 3: Statistically significant difference between self-administered and interview data, but no statistically significant difference between validated and not validated language versions

→ Merging of AFEQT data from validated and not validated language versions and separate analyses of data from both groups (self-administered vs. interview) regarding all further analyses

Scenario 4: No statistically significant difference between self-administered and interview data and no statistically significant difference between validated and not validated language versions

→ Merging of AFEQT data from validated and not validated language versions and merging of data from both groups regarding all further analyses

# 7 Data Handling

This chapter contains instructions for data handling which are generally decisive for derived variable calculations and data presentation.

The basis for time calculations will be the first documented procedure (SAP chapter 7.4.1).

In order to assess the effects of patients lost to follow-up, percentages of dropouts and reason for loss to follow-up will be summarized. In addition, baseline characteristics of patients who were lost to follow-up in comparison to patients with a complete follow-up will be described (SAP chapter 8.6). Patients who withdrawal the PIC/PDRF will be handled according to SAP chapter 6.1.

### 7.1 Definitions

#### Pre-post differences

Pre-post differences in absolute values (also called absolute changes) will always be calculated as post-baseline value minus baseline value.

#### Relative pre-post differences

Relative pre-post differences (also called percent changes) will always be calculated as 100% (post-baseline value minus baseline value) / baseline value.

Pre-post differences will be calculated for the following variables (other can be proposed retrospectively):

**Table 2:** Variables for pre-post differences

| Variables | Pre- value | Post- value | Derived variables |
|---|---|---|---|
| Antiarrhythmic medication<br>Anticoagulation medication<br>Antiplatelets<br>Other cardiovascular medi-<br>cation | Discharge | 12MFU visit/<br>12MFU by<br>phone | Number of patients |
| AFEQT-Score | Baseline | 12MFU/<br>12MFU by<br>phone | Absolute change in AFEQT score |
| AF burden | Baseline | 12MFU visit/<br>12MFU by<br>phone | Absolute change in AF burden [%] |
| EHRA AF symptoms classification | Baseline | 12MFU visit/<br>12MFU by<br>phone | |

# 7.2 Handling data entity types

The CDISC data export is arranged according to the tables in the eCRF (see Data Management Plan). These tables contain data of entities, whose definitions only partially correspond to the entity types processed in statistical analysis. The aim of the analysis is to show the data at patient level.

The following entity types can be used for statistical analysis:

- 1. Patient
- 2. Procedure
- 3. Follow-up
- 4. Adverse Event

#### 7.2.1 Patient data

Data will be analysed showing data on patients level according the eCRF segments enrolment, demographics, medical history, concomitant diseases, diagnostics, medication, hospital discharge, quality of life (AFEQT) and study exit.

#### 7.2.2 Procedural data

Procedure data will be displayed separately according to their chronology. Additional procedures will be shown individually including all procedure details, such as for the first documented procedure. The first documented procedure is the basis for main objective calculations (SAP chapter 8.1). Discharge belonging to procedure: Hospital discharge after an additional procedure. For patients with several procedures, there may be several discharge events, too. All events will be processed and analysed, just as the medications associated with the procedure.

## 7.2.3 Follow-up data

Only unique 12MFU form per patient will be used for analysis. If a General Follow-up visit meets the time window of the 12MFU visits (>351d after procedure), manually data review and selection will be performed. Any FU forms older than 440 days after procedure will not be used for analysis (protocol deviation). For patients with contradictory information in the eCRF the following rules are applied:

- 1. 12 month FU (by phone or visit) is preferred to GFU.
- 2. Events are always kept, even if GFUs are discarded.

The decision on patient level is given in Appendix F.

12MFU visit and 12MFU by phone results will be analysed combined, where variables were recorded in a similar manner (demographics, symptoms, hospitalization, medication). Not combinable information will be shown separately.

General FU (GFU) data will be assigned to the respective time period after first documented procedure:

- 0 to 3 months (1 day =< time between procedure and GFU <= 90 days)
- 3 to 6 months (90 days < time between procedure and GFU <= 180 days)
- 6 to 9 months (180 days < time between procedure and GFU <= 270 days)
- 9 to 12 months (270 days < time between procedure and GFU <= 351 days)

Multiple GFU per patient within one time period will be shown separately in chronological order (i.e. all first GFUs in one time period, all second GFUs in one time period and so on) as descriptive tables.

Number of GFUs per time period and time (days) until GFU during the time period (for each visit per time period) will be shown. Event rates for clinical events (history of AF, reablations and hospitalizations) will be calculated for 3, 6 and 9 months after discharge exactly using appropriate statistical methods.

Predefined time windows for GFU from CIP Version 2.0, Table 7.2 will not be applied.

#### 7.2.4 Adverse Event data

Adverse event data (from AE form) will be listed, ordered and reported by seriousness and relatedness to the procedure. Further adverse event analysis are described in the additional objective of this study (SAP chapter 8 and 8.2). For Adverse event analysis only AEAC adjudicated (SUO form) events will be analysed.

# 7.3 Categorisations

Variable categorisations will be done and displayed for all variables created for subgroup definitions (number of patients treated with PVAC GOLD solely). Following variable categorisations will be also displayed:

- Age by categorisation 1 [years]: <65, 65-74, ≥75</li>
- Age by categorisation 2 [years]: <65, 65-75, >75, 75-80, >80
- Weight [kg]: ≤60, >60
- Body Mass Index [kg/m²]: <18.5, 18.5 to <25, 25 to <30, ≥30 (including WHO obesity classes I-III)</li>
- Number of drinks/day > 10
- HAS-BLED: low, medium, high risk (defined at SAP chapter 7.4.2.1)
- CHA2DS2-VASc: low, medium, high risk (defined at SAP chapter 7.4.2.2)
- Previous ablation (none, 1, ≥ 2)
- Previous surgery for AF (none,  $1, \ge 2$ )
- Hospitalizations due to AF (none,  $1, \ge 2$ )
- INR before ablation (INR≤1, 0.85<INR<1.27, INR≥1)

All other categories will be determined based on the distribution of the respective baseline data. Additional categorisations can be added, if necessary.

#### 7.4 Transformation of Data

## 7.4.1 (Re-)Calculation of derived variables

Body Mass Index [kg/m2]
ROUND (body weight [kg] / (body height [cm] / 100) ^2), .01)

Time to event

For the time to event analysis, the time until the occurrence of an event is presented in days [d] and calculated as follows:

Date of event occurrence – date of first documented procedure

#### Length of stay in rehabilitation [days]

ROUND((Date of discharge - Date of referral), 1)

#### **DAPT** [dichotomous]

Dual antiplatelet therapy: Combination of Aspirin and an P2Y<sub>12</sub> inhibitor (Clopidogrel, Prasugrel or Ticagrelor).

#### **Procedure Timing**

- General time of the procedure = defined and calculated by eCRF
- Time in between vessel access = time of last catheter removal first vessel access
- Lab occupancy time = Time patient left the Catheter Lab Time patient delivered to the Catheter Lab
- PVAC ablation time = Time of last PVAC ablation Time of first PVAC ablation
- MAAC duration = Time of last MAAC ablation Time of first MAAC ablation
- MASC duration = Time of last MASC ablation Time of first MASC ablation

#### 7.4.2 Risk scores

#### 7.4.2.1 HAS-BLED Score

The HAS-BLED Score is based on nine variables which contribute (if fulfilled) to the score by each point:

| Risk Factor / Variable | Points |
|--------------------------------------------------------|--------|
| <u>H</u> ypertension* | 1 |
| <u>A</u> bnormal renal function liver function | 1<br>1 |
| <u>S</u> troke/TIA | 1 |
| <b>B</b> leeding | 1 |
| <u>L</u> abile INR | 1 |
| <b><u>E</u></b> Iderly (> 65) | 1 |
| <b>D</b> rugs (antiplatelets or NSAID) alcohol abuse** | 1<br>1 |

<sup>\*</sup> Hypertension is defined as present, if hypertension is ticked "yes" and/or the systolic BP is ≥ 160mmHg

If one of the variables that is contributing to the HAS-BLED Score is missing, the score is not calculated.

<sup>\*\*</sup> Alcohol abuse is defined as ≥2 drinks per day

The maximum of the HAS-BLED Score is 9 points. A categorisation into low / medium / high risk is given by:

| Range | Risk |
|-----------|--------|
| 0 or 1 | low |
| 2 | medium |
| 3 or more | high |

#### 7.4.2.2 CHA<sub>2</sub>DS<sub>2</sub>-VASc Score

The CHA<sub>2</sub>DS<sub>2</sub>-VASc Score is based on eight variables which contribute (if fulfilled) to the score by each point:

| Risk Factor / Variable | Points |
|---|---|
| Congestive heart failure/LV dysfunction* | 1 |
| <u>H</u> ypertension** | 1 |
| <b>A</b> ge > 75 | 2 |
| <u>D</u> iabetes Mellitus | 1 |
| $\underline{\mathbf{S}}$ troke or TIA or thromboembolic event | 2 |
| $\underline{\mathbf{V}}$ ascular disease (prior myocardial infarction, peripheral artery disease, or complex aortic plaque) | 1 |
| <b>A</b> ge 65 – 74 y | 1 |
| <u>S</u> ex <u>c</u> ategory (female gender) | 1 |

<sup>\*</sup> Congestive heart failure / LV dysfunction is defined as present, if chronic heart failure is ticked "yes"

If one of the variables that is contributing to the CHA<sub>2</sub>DS<sub>2</sub>-VASc Score is missing, the score is not calculated.

The maximum of the  $CHA_2DS_2$ -VASc Score is 9 points. A categorisation into low / medium / high risk is given by:

| Range | Risk |
|-----------|--------|
| 0 | low |
| 1 | medium |
| 2 or more | high |

## 7.4.3 Scoring of questionnaire data (AFEQT)

Symptom subscale score

<sup>\*\*</sup> Hypertension is defined as present, if hypertension is ticked "yes"

In a first step, the levels of the 7 answer categories (equal to the order of appearance) for the 4 questions contributing to the Symptom subscale (i.e. questions 1, 2, 3, 4) are coded as follows:

| level 1 (not at all bothered<br>OR I did not have this symptom) | <b>→</b> 1 |
|---|---|
| level 2 (hardly bothered) | $\rightarrow$ 2 |
| level 3 (a little bothered) | <b>→</b> 3 |
| level 4 (moderately bothered) | $\rightarrow 4$ |
| level 5 (quite a bit bothered) | <b>→</b> 5 |
| level 6 (very bothered) | <b>→</b> 6 |
| level 7 (extremely bothered) | <b>→</b> 7 |

In a second step, using the assigned values the Symptom subscale is calculated as follows:

#### Daily Activities subscale score

In a first step, the levels of the 7 answer categories (equal to the order of appearance) for the 8 questions contributing to the Daily Activities subscale (i.e. questions 5, 6, 7, 8, 9, 10, 11, 12) are coded as follows:

#### (a) Questions 5 and 6:

| level 1 (not at all limited) | $\rightarrow 1$ |
|---------------------------------|-----------------|
| level 2 (hardly limited) | $\rightarrow$ 2 |
| level 3 (a little limited) | $\rightarrow$ 3 |
| level 4 (moderately limited) | $\rightarrow 4$ |
| level 5 (quite a bit limited) | $\rightarrow$ 5 |
| level 6 (very limited) | <b>→</b> 6 |
| level 7 (extremely limited) | $\rightarrow$ 7 |
| (b) Questions 7 to 12: | |
| level 1 (no difficulty at all) | $\rightarrow 1$ |
| level 2 (hardly any difficulty) | $\rightarrow$ 2 |
| level 3 (a little difficulty) | <b>→</b> 3 |
| level 4 (moderate difficulty) | $\rightarrow 4$ |

| level 5 (quite a bit of difficulty) | $\rightarrow$ 5 |
|-------------------------------------|-----------------|
| level 6 (a lot of difficulty) | <b>→</b> 6 |
| level 7 (extreme difficulty) | <b>→</b> 7 |

In a second step, using the assigned values the Daily Acivities subscale is calculated as follows:

#### Treatment Concern subscale score

In a first step, the levels of the 7 answer categories (equal to the order of appearance) for the 6 questions contributing to the Symptom subscale (i.e. questions 13, 14, 15, 16, 17, 18) are coded as follows:

| level 1 (not at all bothered | $\rightarrow 1$ |
|--------------------------------|-----------------|
| level 2 (hardly bothered) | $\rightarrow$ 2 |
| level 3 (a little bothered) | <b>→</b> 3 |
| level 4 (moderately bothered) | $\rightarrow 4$ |
| level 5 (quite a bit bothered) | <b>→</b> 5 |
| level 6 (very bothered) | <b>→</b> 6 |
| level 7 (extremely bothered) | <b>→</b> 7 |

In a second step, using the assigned values the Treatment Concern subscale is calculated as follows:

#### Treatment Satisfaction subscale score

In a first step, the levels of the 7 answer categories (equal to the order of appearance) for the 2 questions contributing to the Symptom subscale (i.e. questions 19, 20) are coded as follows:

| level 1 (extremely satisfied) | $\rightarrow 1$ |
|-------------------------------------------------|-----------------|
| level 2 (very satisfied) | $\rightarrow$ 2 |
| level 3 (somewhat satisfied) | $\rightarrow$ 3 |
| level 4 (mixed with satisfied and dissatisfied) | $\rightarrow 4$ |

| level 5 (somewhat dissatisfied) | $\rightarrow 5$ |
|----------------------------------|-----------------|
| level 6 (very dissatisfied) | <b>→</b> 6 |
| level 7 (extremely dissatisfied) | <b>→</b> 7 |

In a second step, using the assigned values the Treatment Satisfaction subscale is calculated as follows:

#### Overall AFEQT score

In a first step, the levels of the 7 answer categories (equal to the order of appearance) for the 20 questions contributing to the Symptom subscale (i.e. questions 1 to 20) are coded as follows:

 $\rightarrow 1$ 

#### (a) Questions 1 to 4:

level 1 (not at all bothered

| OR I did not have this symptom) | |
|---------------------------------|-----------------|
| level 2 (hardly bothered) | $\rightarrow$ 2 |
| level 3 (a little bothered) | $\rightarrow$ 3 |
| level 4 (moderately bothered) | $\rightarrow 4$ |
| level 5 (quite a bit bothered) | $\rightarrow$ 5 |
| level 6 (very bothered) | $\rightarrow$ 6 |
| level 7 (extremely bothered) | $\rightarrow$ 7 |
| (b) Questions 5 to 6: | |
| level 1 (not at all limited) | $\rightarrow 1$ |
| level 2 (hardly limited) | $\rightarrow 2$ |
| level 3 (a little limited) | $\rightarrow$ 3 |
| level 4 (moderately limited) | $\rightarrow 4$ |
| level 5 (quite a bit limited) | $\rightarrow$ 5 |
| level 6 (very limited) | <b>→</b> 6 |
| level 7 (extremely limited) | $\rightarrow$ 7 |
| (b) Questions 7 to 12: | |
| level 1 (no difficulty at all) | $\rightarrow 1$ |

| level 2 (hardly any difficulty) | $\rightarrow$ 2 |
|-------------------------------------------------|-----------------|
| level 3 (a little difficulty) | <b>→</b> 3 |
| level 4 (moderate difficulty) | $\rightarrow 4$ |
| level 5 (quite a bit of difficulty) | <b>→</b> 5 |
| level 6 (a lot of difficulty) | <b>→</b> 6 |
| level 7 (extreme difficulty) | <b>→</b> 7 |
| (c) Questions 13 to 18: | |
| level 1 (not at all bothered | $\rightarrow 1$ |
| level 2 (hardly bothered) | $\rightarrow$ 2 |
| level 3 (a little bothered) | <b>→</b> 3 |
| level 4 (moderately bothered) | $\rightarrow 4$ |
| level 5 (quite a bit bothered) | $\rightarrow 5$ |
| level 6 (very bothered) | <b>→</b> 6 |
| level 7 (extremely bothered) | <b>→</b> 7 |
| (d) Questions 19 to 20: | |
| level 1 (extremely satisfied) | $\rightarrow 1$ |
| level 2 (very satisfied) | $\rightarrow 2$ |
| level 3 (somewhat satisfied) | <b>→</b> 3 |
| level 4 (mixed with satisfied and dissatisfied) | $\rightarrow 4$ |
| level 5 (somewhat dissatisfied) | <b>→</b> 5 |
| level 6 (very dissatisfied) | <b>→</b> 6 |
| level 7 (extremely dissatisfied) | <b>→</b> 7 |

In a second step, using the assigned values the Overall AFEQT score is calculated as follows:

100 - (sum of severity for all questions answered - number of questions answered) X 100 (total number questions answered X 6)

# 7.5 Replacement of Data

## 7.5.1 Replacement of missing values

All reasonable attempts will be undertaken to ensure completeness of data collection in this registry. Before database lock, as many queries as possible will be cleared. If Note to Files arises after database closure (baseline data base lock or final database lock) that relate to data analysis, the data is changed accordingly for analysis.

According to the Clinical Investigational Plan, missing values will not be replaced for any of the parameters in the statistical analysis. Only observed cases will be evaluated.

#### 7.5.2 Replacement of outliers

In general, outliers are evaluated as reported. In the event of highly implausible values (in the sense of extreme outliers) documented in the database after completion of data validation the following approach is used:

For some baseline variables (e.g. age, weight, height) as well as for vital signs so-called plausibility ranges will be defined (Table 3).

Observed values that are not within these ranges are set to missing within the analysis datasets. The intention of these ranges is to set them as wide as possible, so that only values that are obviously impossible (e.g. age of 150 years or systolic blood pressure of 20 mmHg) are set to missing. Borderline values confirmed by the investigator within a query will not be set to missing.

The definition of the ranges is always set in consultation with a medical expert. An appropriate documentation of the implausibility ranges is given in the following table of this SAP according to the ranges in the Data Validation Plan.

**Table 3: Ranges** 

| Value | Range |
|--------------------------------------------------|------------------|
| Height | 90 - 250 cm |
| Weight | 30 - 500 kg |
| BMI (automatically calculated) | 15 - 40 |
| Age | 18 - 120 years |
| Catheter PV cryo ablation - Total no. | 1 - 4 |
| Catheter PV rf ablation - Total no. | 1 - 4 |
| Catheter PV 3D RF ablation - Total no. | 1 - 4 |
| Number of pharmalogical cardioversions | 1 - 99 Total no. |
| Number of electrical cardioversions | 1 - 99 Total no. |
| Number of admissions | 1 - 9 Total no. |
| Number of drinks/day | 5 - 99 |
| AF burden (optional) | 0 - 100 % |
| Documented LVEF | 15 - 70 % |
| Documented anteroposterior left aterial diameter | 0 - 100 mm |
| INR value | 0,5 - 9 |

| General time of the procedure | 30 - 300 min |
|----------------------------------------|------------------|
| LSPV | 0 - 40 no. |
| LIPV | 0 - 40 no. |
| LCPV | 0 - 40 no. |
| RSPV | 0 - 40 no. |
| RIPV | 0 - 40 no. |
| RMPV | 0 - 40 no. |
| Other accesery vein | 0 - 40 no. |
| Number of pharmalogical cardioversions | 1 - 20 Total no. |
| Number of electrical cardioversions | 1 - 20 Total no. |
| Documented LVEF | 0 - 100 % |
| Number of pharmalogical cardioversions | 1 - 99 Total no. |
| Number of electrical cardioversions | 1 - 99 Total no. |
| AF burden | 0 - 100 % |

#### 7.6 Self-Evident Corrections

Self-evident corrections will not be implemented in the raw data but on basis of the analysis data sets. They are described in the Data Validation Plan.

# **8** Descriptive Statistics

This section describes the most relevant parts of the statistical analyses planned for this registry. All planned statistical methods will be described in detail in the Statistical Analysis Plan, which should be finalized prior to interim analysis and need to be finalized prior final analysis.

In general, this registry is intended to collect data under real life conditions. The statistical analysis will be performed in explorative and descriptive manner, i.e. no pre-specified hypothesis testing.

All variables collected in the CRF as well as the data obtained from the QoL assessments and all derived parameters will be used in the statistical analysis.

Binary, categorical, and ordinal parameters will be summarized by means of absolute and percentage numbers within the various categories.

Continuous data will be summarized by means of standard statistics, i.e. number of available data, number of missing data, mean, standard deviation, minimum, median, maximum, 5<sup>th</sup> and 95<sup>th</sup> percentile, lower and upper quartile (see SAP Appendix A).

Time-to-event data is planned to be analysed via a Cox proportional hazard regression model presenting hazard ratios and the corresponding 95% CI. In addition, Kaplan-Meier

curves may be presented for the time-to-event data. Two-sided 95%-CI will be presented for important parameters, but should be interpreted in an exploratory descriptive way. No formal statistical tests are planned within the statistical analysis. Event rates will be calculated for 3, 6, 9 and 12 months after first documented procedure and may be displayed graphically.

To measure statistical differences in continuous or dichotomous/ multinomial variables between baseline and 12 month FU non-parametric (e.g. Friedman's Chi-Square Test, McNemar's Test) will be utilized. The test is only performed if the variable is not missing at admission and discharge.

A biometrical report including descriptive statistics of all relevant documented parameters will be generated for the overall patient population as well as for each participating country (SAP chapter 8.7). Depending on the variable(s) of interest, additional selection criteria for subjects (e.g. subgroup analyses) considered in specific analyses may be used, if considered useful during the statistical analysis (SAP chapter 8.6).

Any change to the data analysis methods described in the CIP will require an amendment only if it changes main and additional objectives of the CIP. Any other changes to the data analysis methods described in the CIP, and the justification for making the change, will be described in the clinical study report<sup>1</sup>.

In order to assess the effects of patients lost to follow-up, percentages of dropouts and reason for loss to follow-up will be summarized. In addition, baseline characteristics of patients who were lost to follow-up in comparison to patients with a complete follow-up will be described.

Additionally, adequate graphs (e.g. bar charts, box-whisker plots) may be presented to summarize the results for some parameters. Further descriptive statistical analyses will be carried out, e.g. correlation analysis (SAP chapter 8.8).

## 8.1 Statistical analyses for the main objective

#### 8.1.1 Estimate Phased RFA 12 month success rate

Success rate estimated as the time to first AF re-occurrence event from the first documented procedure. Data about AF events will be collected since the first documented procedure, including 90 days of the "blanking period" and closes at 12 months FU. If no AF events occur during the follow-up period (considering the "blanking period") up to 12 (+2) months, the case is considered to be "event-free". Calculations will be done for exact 12 months (351 days) after first documented procedure.

Main objective will be calculated for the BAS, FAS and EFAS (see chapter 4 and Appendix B). A successful first documented procedure (successfulness by PVI confirmation) is the basis to calculate the main objective. Patients with a procedure during the "blanking

<sup>&</sup>lt;sup>1</sup> in the service agreement #2 refers to the final report, which is one and the same document for this study

period" of 90 days after first documented procedure will be excluded from main objective calculations.

Predefined AF re-occurrence definition from CIP Version 2.0 will not be applied to calculate the main objective. Further analysis might be used to estimate Phased RFA success rate considering (re-)occurring left Afl events.

AF re-occurrence event defined as:

- AF pharmacological and/or electrical CV
- o AF more the 30 sec on ECG/EGM
- o AF less than 30 sec in combination with AF symptoms
- Re-ablations for AF

For this analysis adjudicated AE data and coded AE data (free text fields) will be used. AF re-occurrence event rate will be estimated with and without the use of antiarrhythmic drugs at time of the 12 month follow-up. AF re-occurrence rates will be calculated for patients from BAS and FAS (Appendix B) which need to have a signed 12 month FU / 12 month FU by phone form by definition. AF re-occurrence is defined as the first event of AF re-occurrence event and their related date information based on the following eCRF forms and data fields:

| eCRF field | Related date field | <b>Related FID's</b><br>annotated eCRF (V1.3,<br>V1.4) |
|---|---|---|
| Reason for visit: AF re-occurrence | Date of visit | F11000050<br>F11000010 |
| Re-ablation reason: Due to AF-<br>occurrence | Date of visit | F11000070<br>F11000010 |
| History of arrhythmias since last visit: AF | Date of first occur-<br>rence | F12000012<br>F12000050 |
| History of arrhythmias since last visit: Reablation for AF | Date of re-ablation<br>for AF | F12000060<br>F12000070 |
| CVD hospitalizations during last visit: AF | Date of first admission | F15000020<br>F15000030 |

Table 4: Main objective variables at 12MFU / General FU form

**Table 5:** Main objective variables at 12MFU by phone form

| eCRF Field | Related date<br>field | Related FID's<br>annotated eCRF (V1.3,<br>V1.4) |
|---|---|---|
| History of arrhythmias since last visit: AF | Date of first occur-<br>rence | F13000010<br>F12000050 |
| History of arrhythmias since last visit:<br>Re-ablation for AF | Date of re-ablation<br>for AF | F12000060<br>F12000220 |
| CVD hospitalizations during last visit:<br>AF | Date of first ad-<br>mission | F15000010<br>F15000020_1<br>F15000030 |

**Table 6:** Main objective variables at AE form

| eCRF Field | Related date field | Related FID's<br>annotated eCRF (V1.3,<br>V1.4) |
|---|---|---|
| Other diagnostics: ~"AF" | Date of AE | F31000010_88<br>F30000090<br>F30000010 |

## 8.1.2 Methodology for analysing the main objective

Any AF re-occurrence event (Tables 5, 6 and 7) during the "blanking period" will be not be considered. "Blanking period" starts with the day of the first documented procedure and ends at exact 90 days. The first documented date of AF re-occurrence will be set as the event date. "Blanking period" for patients with additional procedure(s) at any time will not be started newly, they will be considered as "not-event free" at time of the first additional procedure.

Freedom from AF re-occurrence at 12 months will be estimated using Kaplan-Meier methods (time-to-first-event-analysis). A point estimate at the date of 12MFU post first documented procedure will be presented. Standard error will be approximated using
Greenwood's formula, and a two-sided 95% log-log confidence interval will be presented. For patients without a reported AF re-occurrence event, those patients will be censored. In this case, the right-censoring time will be set to the last study contact date. Main objective Kaplan-Meier estimation results will be displayed in percentages at 12 months (351 days) after first documented procedure. Estimated AF re-occurrence rates by month (at the end of month 3 to 11 after first documented-procedure) will be calculated and displayed as well. For group comparisons Log-Rank test will be applied. Also, Hazard ratios and 95% confidence intervals will be shown (for group comparisons, please see SAP chapter 8.6). For Kaplan-Meier estimation, numbers at risk will be displayed for reasonable points in time.

Re-occurrence of AF during 12 months (considering the "blanking period") will also be analysed via Cox proportional hazard regression model presenting hazard ratios and the corresponding 95% CI. Independent variables will be determined by Phased RFA procedure experts or physicians. Cox modelling for AF re-occurrence will be done for all predefined subgroups (FAS patients) where the analysis scope is the 12 month outcome (SAP chapter 8.6.1). Further Cox modelling (e.g. for multiple AF events) may be applied.

#### 8.2 Statistical analyses for additional objective

#### 8.2.1 Estimate Phased RFA procedure safety

Major procedure related complications include vascular complications secondary to venous access, cardiac tamponade, embolic stroke, esophageal injury, phrenic nerve injury, PV stenosis, reentrant tachycardia arrhythmias arising from ablations, mainly left Afl.

Adverse events (AE) including their relatedness to the respective procedure, are documented starting from the first documented procedure until the 12 month FU. For this analysis only adjudicated AE data (SUO form) and coded AE data (from free text fields) will be used. In addition, TIA/Stroke events will be taken from general FU forms to calculate procedure safety. Analysis will be performed at 30 days and at 12 months after procedure.

If no adverse event was documented within the 12 month FU period, the patient or the procedure is considered to be "free of AE". AEs are documented in the AE form, whereby distinctions in relatedness to which procedure (index phased RFA, repeated phased RFA or phased RFA re-ablation) will be made. Phased RFA procedure relatedness will also be taken from the AE form (Relatedness to Phased RFA procedure = related). The documented date of the AE will be used to set the point in time. For analysis purposes, phased RFA procedure safety will be calculated for first documented procedures (on procedure and patient level), separated for additional procedures (on procedure level) and for patients with additional procedures (on patient level).

Procedure safety will be calculated for procedures that have been carried out (number of RF applications per patient > 0) and disregarding procedure successfulness. This study objective will be calculated for the BAS and the FAS (Appendix B) for patients with signed eCRF.

Further analysis might be performed, e.g. procedure safety for using PVAC GOLD solely or not PVAC GOLD solely (using other catheter or using adjunctive devices).

 Table 7: Procedure safety variables at AE form

| AE due to definition | eCRF field: AE description | Related FID's<br>annotated eCRF<br>(V1.3, V1.4) |
|---|---|---|
| Vascular access complication | Vascular access complication | F31000010_6 |
| Cardiac tamponade | Pericardial damage | F31000010_8 |
| Stroke | Stroke | F31000010_2 |
| Esophageal injury | Atrioesophageal damage | F31000010_9 |
| Phrenic nerve injury | Phrenic nerve damage | F31000010_7 |
| PV stenosis | PV stenosis Symptomatic or Asymptomatic of diameter of stenosis ≤ 50% or >50% or NA | F31000010_1<br>F31000030 |
| Re-entrant tachycardia ar-<br>rhythmias arising from abla-<br>tions | Other (diagnosis)<br>Description field | F31000010_88<br>F31000090 |
| Mainly left Afl | Left Afl | F31000010_11 |
| Other diagnostics: text complies to AEs above, text will be coded | Free text field | F31000010_88<br>F30000090<br>F30000010 |

**Table 8:** Procedure safety variables at FU form

| AE due to definition | eCRF field: AE description | Related FID's<br>annotated eCRF<br>(V1.3, V1.4) |
|---|---|---|
| Stroke | • TIA/Stroke | F15000140<br>F15000150 |

#### 8.2.2 Methodology for analysing the procedure safety

The number of patients with reported device and procedure related events will be summarized as a binomial variables for each event and combined; number and percentage of events and patients with events (up to 12 month after first documented procedure). Additionally, Kaplan-Meier estimations (time-to-first-event analysis) will be used to summary the timing of the occurrence of safety events through 30 days and 12 months (351 days) after first documented procedure. Time from onset to resolution of events will also be presented. Further strata may be applied for analysis (e.g. reason for ablation: index, repeated, re-ablation, left Afl).

#### 8.3 Statistical analyses for ancillary objectives

According to Appendix B, these analyses will be performed for the Baseline Analysis Set and Full Analysis Set. If not described otherwise, ancillary objectives will be analysed using methods of descriptive statistics (SAP chapter 8).

#### 8.3.1 Characterize the acute procedural success rate

Success rates will be calculated for all documented procedures combined (patient level). Also, procedure success rates will be provided for first documented procedures, additional procedures, regular cases and training cases, separately. Success rates will also be shown per vein.

Success will be calculated for procedures that have been attempted (number if RF applications per patient > 0). Success rates will be provided for PVAC GOLD solely procedures (ancillary objective) and additionally for not PVAC GOLD solely procedures (using other catheter and/or using adjunctive devices).

If RF applications per patient, consumables (Phased RFA catheters used), successfulness and PV confirmation (exit or entrance block) was not verified for the procedure, the data will not be used for analysis. Consumables and procedure success will be taken from the procedure form. Relatedness of Phased RFA will be taken from AE form.

The procedure is considered successful if:

- Procedure attempt was not declined due to technical issues related to Phased RFA system and
- Only PVAC catheter(s) used to achieve PVI and
- All accessible PVs were isolated (entrance and/or exit block confirmation per vein)

This combined endpoint (variables linked via "and operation") is applicable, if all conditions are available and complied.

Because of different procedure forms (eCRF V1.3 and eCRF V1.4), PVI achievement by PVAC GOLD only is assumed for patients documented by eCRF V1.3 as follows:

- [F21000010] Phased RFA catheter used: only PVAC GOLD is ticked, and
- [F22000010] to [F22000060] PVI confirmation: exit block and/or entrance block are ticked, and
- [F20001000] Number of RF applications per patient > 0

Unsuccessfulness per vein is considered, if the vein is not isolated or not verified. Percentages for success will be shown per vein for patients treated with PVAC GOLD solely. Precondition is that the number of RF applications per patient is greater than zero.

PVI achievement by PVAC GOLD only is defined for patients documented by eCRF V1.4 as follows:

- [F21000010] Phased RFA catheter used: only PVAC GOLD is ticked, and
- [F22000062] Where all PVs isolated at the end of the procedure = yes, and
- [F22000066] Where all PVs isolated by using PVAC only = yes, and
- [F21000010] Number of RF applications per patient > 0

Unsuccessfulness per vein is considered, if the vein is not isolated or not verified. Percentages for success will be shown per vein for patients treated with PVAC GOLD, all PVs were isolated at the end of the procedure = no and all PVs isolated by using PVAC only = no.

**Table 9:** Procedure success variables from Procedure and AE form

| Objective section | Definition (used variables) | Related FID's |
|---|---|---|
| | | annotated eCRF |
| | | (V1.3, V1.4) |
| Procedure attempt was not de- | Procedure form: | F20000010 |
| clined due to technical issues re- | Date of procedure | F22000180 |
| lated to Phased RFA system | Phased RFA procedure successful? | F22000190 |
| | No – Due to AE | |
| | AE form: | |
| | Date of AE | |
| | Was the event related to technical | F30000010 |
| | issues?* | F30000070 |
| | Related/Possibly related | CD5) /4 2 4 /4 /4 |
| Only PVAC catheter(s) used to | Procedure form: | eCRFV1.3/V1.4 |
| achieve PVI | Phased RFA catheters used PVAC GOLD (solely) | F21000010 |
| | Number of RF applications per patient > 0 | F20001000 |
| | ' ' | eCRFV1.4 only |
| | Were all PVs isolated at the end of the procedure | F22000062 |
| | Were all PVs isolated by using only PVAC | F22000066 |

| All accessible PVs were isolated | Were all accessible PVs isolated at | eCRFV1.3/V1.4 |
|---|---|---|
| (entrance and/or exit block con- | the end of the procedure entrance | F22000010 |
| firmation per vein) | block and/or exit block | F22000020 |
| , and the second | Exit block and/or | F22000030 |
| | Entrance block | F22000040 |
| | | F22000050 |
| | | F22000060 |

<sup>\*</sup> Precondition: If the documented AE is related to technical issues with Phased RFA system components, the date of the latest procedure must be ≤ date of the AE. For patients with more > 1 procedure, the latest procedure will be the related procedure.

#### 8.3.1.1 Methodology for analysing the acute procedural success rate

Acute procedural success rate will be reported as frequency and percentages. Acute procedural success rate by patients will be calculated as number of patients with acute procedural success divided by number of patients with an attempted Phased RFA procedure. Acute procedural success rate by vein will be calculated as number of veins with electrical isolation verified divided by number of veins attempted with Phased RFA. 95% confidence intervals will be calculated using Fisher's exact method.

#### 8.3.2 Assess Phased RFA efficiency

Phased RFA efficacy data will be shown for all documented procedures combined (patient level). Also, phased RFA efficacy will be provided for first documented procedures, additional procedures, regular cases and training cases, separately.

The parameters to measure the efficiency:

- Procedure duration
- Laboratory occupancy duration
- Fluoroscopy time
- Phased RFA consumables used
- Adjunctive devices (mapping or navigation systems)

**Table 10:** Phased RFA efficiency variables from procedure form

| Objective section | Objective section Definition (used variables) | |
|---|---|---|
| | | annotated CRF<br>(V1.3, V1.4) |
| Procedure duration | General time of the procedure | F20000611 |
| Laboratory occupancy duration | Time patient delivered to the Catheter Lab | F20000420 |
| | Time patient left the Catheter Lab | F20000610 |
| Fluoroscopy time | Total fluoroscopy time | F20000620 |
| Phased RFA consumables used | General number of catheters used | F21000005 |
| | Phased RFA catheters used | F21000010 |
| | Other (free text field) | F21000020 |
| Adjunctive devices (mapping or navigation systems) | Adjunctive devices used during the procedure | F21000040 |
| | Other (free text field) | F21000050 |

Phased RFA efficiency will be analysed for all implemented procedures only (number if RF applications per patient > 0). Time data will be shown for PVAC GOLD solely and using different catheters or adjunctive devices. Additionally, it will be distinguished between reasons of ablation (index, repeated, re-ablation, left Afl).

#### 8.3.3 Characterize the peri-procedural anticoagulation therapy

Peri-procedural anticoagulation therapy data will be shown for all documented procedures combined (patient level). Also, peri-procedural anticoagulation therapy will be provided for first documented procedures, additional procedures, regular cases and training cases, separately.

The parameters of interest:

- Activated clotting time (ACT) during the procedure
- Peri-procedural INR
- Oral anticoagulant therapy/LMWN before, during and after the procedure
- TIA/stroke related to study Phased RFA procedure

**Table 11:** Peri-procedural anticoagulation therapy variables from baseline, procedure and AE form

| Objective section | Definition (used variables) | Related FID's |
|---|---|---|
| , | , | annotated eCRF<br>(V1.3, V1.4) |
| Activated clotting time (ACT) during the procedure | Highest ACT during procedure<br>Lowest ACT during procedure | F20000300<br>F20000320 |
| Peri-procedural INR | Latest measured INR<br>INR value<br>Date of INR test | F20000260<br>F20000270<br>F20000280 |
| Oral anticoagulant therapy/LMWN before, during and after the procedure | Procedure form: Was oral anticoagulant discontinued before the procedure | F20000210 |
| | How many hours prior to procedure Was LMWH administered before the | F20000220 |
| | procedure Instead of oral Anticoagulants | F20000230 |
| | In addition to the oral anticoagulants | F20000240 |
| | Baseline form (prior procedure):<br>Anticoagulation Medication<br>Specify (free text field) | F20000250 |
| | Procedure form (after procedure): Was anticoagulation continued after the procedure How long after procedure | F17500100<br>F17500120 |
| | Procedure form (after procedure/at discharge): | F23000060 |
| | Anticoagulation Medication<br>Specify (free text field) | F23000070 |
| | | F19500100<br>F19500120 |

| TIA/stroke related to s | study | Procedure form: | F20000010 |
|---|---|---|---|
| Phased RFA procedure | - | Date of procedure | F22000180 |
| · | | Phased RFA procedure successful? | F22000190 |
| | | No – Due to AE | |
| | | AE form:<br>Date of AE | |
| | | | F30000010 |
| | | | F31000010_2 |
| | | | F31000010_3 |

## 8.3.4 Describe single catheter PVAC GOLD utilization in persistent AF

Single PVAC GOLD utilization data will be shown for all documented procedures combined (patient level). Also, single PVAC GOLD utilization will be provided for first documented procedures, additional procedures, regular cases and training cases, separately.

Single catheter PVAC GOLD utilization means here, that only PVAC GOLD was used during the procedure, regardless of using sheaths. No adjunctive devices were used. For this ancillary objective, only patients with persistent AF will be analysed.

The parameters of interest are:

- Phased RFA catheters used during the procedure
- Indication for Phased RFA
- Location of linear lesions or substrate modifications
- Atrial CV
- AF/ left Afl recorded on ECG/EGM
- AF re-ablations

**Table 12:** PVAC GOLD utilization variables from baseline and procedure form

| Objective section | Definition (used variables) | Related FID's |
|---|---|---|
| | , | annotated eCRF<br>(V1.3, V1.4) |
| Phased RFA catheters used during the procedure | General number of catheters used Phased RFA catheters used | F21000005 |
| | Other (free text field) | F21000010<br>F21000020 |
| 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 | From procedure form | 540000440 |
| Indication for Phased RFA | Indication to schedule Phased<br>RFA (AF type) | F10000110 |
| | If "Persistent AF" | F10000113 |
| | From baseline form | |
| Location of linear lesions or substrate modifications | Were any non-<br>PVI lesions performed | F20001010 |
| | Substrate Modification = Lines | F20001040 |
| | Location | F20001020 |
| | From procedure form | |

| Atrial CV | Cardioversion(s) for AF in the last 12 months | F13000710 |
|-----------|-----------------------------------------------|-----------|
| | Latest date of CV(s) | F13000720 |
| | specify CV | F13000740 |
| | | F13000750 |
| | | F13000770 |
| | From baseline form | |

#### 8.3.5 Evaluate QoL (AFEQT) dynamic at 12 month FU

Quality of Life analysis will be done for all available subjects. Therefore, completed AFEQT questionnaire at baseline and at 12 month FU will be used. With it, single scales and AFEQT score will be analysed at baseline and at 12 months. Also, absolute and relative differences in AFEQT score between baseline and 12 months will be displayed. Score calculations are described in SAP chapter 7.4.3, rules for analysis in SAP chapter 6.3.

#### 8.4 Interim analysis

Interim analysis (see CIP Version 2.0), based on study data reported prior to the final report, may be completed and utilized for publication. After documenting all intended first documented procedures and pass the query solving process for baseline data, interim database lock will be used to set a locked data set for this analysis. Analysis sets, analysis tables and predefined comparison groups for interim analysis are displayed in Appendix B and D. Ancillary objectives (SAP chapter 8.3.1 to 8.3.4) will be calculated for this data status. Besides, all other parameters from baseline and first documented procedure will be shown. For details see Appendix B. Data analysis will be in descriptive manner. No adjustments for alpha are necessary as no hypotheses are being tested.

#### 8.5 Final analysis

At the end of this study and after the final data base lock, final tables including study objectives (Appendix B), subgroup analysis, comparison group analysis, graphical analysis and benchmark analysis will be performed. Data analysis will be in descriptive manner. No adjustments for alpha are necessary as no hypotheses are being tested.

#### 8.6 Analysis of group comparisons and subgroups

To evaluate special subjects, predefined subgroup analysis and predefined group comparisons will be performed. Subgroup and group comparisons will be done at the end of this study. If needed, further analysis can be carried out.

#### 8.6.1 Analysis of subgroups

Descriptive subgroup reports will be listed in Appendix C.

#### 8.6.2 Analysis of comparison groups

Group comparison will be provided including non-parametric statistical tests and odds ratios with 95% CI (two-group comparison) for all parameters. In Appendix D descriptive reports are listed.

#### 8.7 Benchmark reports

The benchmark reports are a comparison of one single unit (site or country) to the entire group of all other participating units. These benchmark reports are designed to be used as quality control for the participating sites and to describe country differences. Benchmark reports will be provided for:

- Participating site vs. all other sites
- Participating country vs. all other countries

The BAS will be the analysis population. Statistical reports (descriptive statistics) will be provided including all parameters from Baseline, First documented procedure, Additional procedure, GFU and 12MFU, but due to data protection no data from the Adverse Event form. The benchmark reports will be listed in tabular form and, depending on the variable type, the statistical output will include numbers and percentages, mean  $\pm$  SD, Odds ratio with 95% CI for all available parameters.

#### 8.8 Graphical analysis

Graphical analysis will be provided for final analysis. The graphs will be created using SAS. Predefined graphical analysis will be done for the following topics and strata. Additional graphical analyses can be carried out after database closure.

 Table 13: Predefined graphical analysis

| Target variable | Analysis method | Patients set or strata |
|---|---|---|
| Main objective: AF re-occurrence by study definition during 12 months Additional analysis: | Kaplan-Meier estimation<br>(time-to-first-event) | <ul><li>BAS, FAS, EFAS</li><li>AF type</li></ul> |
| AF re-occurrence with and without considering the "blanking period" of 90 days | | |
| AF re-occurrence up to 14 month (end of FU period) after first documented procedure | | |
| Additional objective: Phased RFA procedure safety | Kaplan-Meier estimation<br>(time-to-first-event) | <ul> <li>FAS</li> <li>Reason for ablation:<br/>index, repeated, re-ab-<br/>lation, left Afl</li> </ul> |
| Anticoagulation medication before /during/ after/ at 12months FU | Graphical (stacked) bar<br>analysis | <ul><li>FAS, EFAS</li><li>LAAO implantation</li></ul> |
| Analysis of procedure time by • Site • Operator | Box-whisker plots | • FAS, EFAS |
| Correlation between Anticoagulation and INR ACT Stroke | Suitable correlation methods | • FAS |
| Correlation between AF re-occurrence and BMI Age | Suitable correlation methods | BAS, FAS, EFAS |
| COX regression analysis (SAP chapter 8.1.2) | Forest plot (for HR + CI) | • FAS, EFAS |
| Analysis of DAP - by site | Box-whisker plots | • BAS |

#### 9 References

Camm AJ, Lip GYH, De Caterina R, Savelieva I, Atar D, Hohnloser SH, et al. 2012 focused update of the ESC Guidelines for the management of atrial fibrillation. Eur Heart J. 2012 Nov 1;33(21):2719–47.

Lip GY, Nieuwlaat R, Pisters R, Lane DA, Crijns HJ. Refining clinical risk stratification for predicting stroke and thromboembolism in atrial fibrillation using a novel risk factor-based approach: the Euro Heart Survey on Atrial Fibrillation. Chest 2010;137:263–272.

Pisters R, Lane DA, Nieuwlaat R, de Vos CB, Crijns HJ, Lip GY. A novel user-friendly score (HAS-BLED) to assess 1-year risk of major bleeding in patients with atrial fibrillation: the Euro Heart Survey. Chest 2010;138:1093–1100.

### **Appendix A: Table specifications (examples)**

Table specification for analysis tables (numbers, metric and dichotomous variables)

| Variable | Specification | Format | Nominator<br>(if applicable) | Denominator<br>(if applicable) |
|---|---|---|---|---|
| Number of patients in APS | All patients that met the criteria of the APS | Integer | | |
| Age | | None | | |
| Mean ± SD, N | mean ± standard deviation (format:<br>2 decimal places), number of pa-<br>tients with age values | 2 decimal places,<br>Integer | | |
| Median (Q1-Q3) | median and interquartile range in brackets (format: 2 decimal places) | 2 decimal places | | |
| 5th and 95th Percentile | median and interquartile range in brackets (format: 2 decimal places) | 2 decimal places | | |
| Min, Max | minimal and maximal value (format: 2 decimal places) | 2 decimal places | | |
| Male gender | percentage of male patients | 2 decimal places | male patients | all patients with gen-<br>der information |

# Appendix B: Analysis tables, Study objectives and Analysis sets

| eCRF<br>SEGMENTS | eCRF CHAPTERS/<br>ANALYSIS TABLES | STUDY<br>OBJECTIVES | ANALYSIS SETS<br>FOR INTERIM<br>ANALYSIS | ANALYSIS SETS<br>FOR FINAL<br>ANALYSIS |
|---|---|---|---|---|
| BASELINE | Enrolment | | APS, BAS | APS, BAS, FAS,<br>EFAS |
| | Indication/Admission | | APS, BAS | APS, BAS, FAS,<br>EFAS |
| | Demographics | | BAS | BAS, FAS, EFAS |
| | History of CVD | | BAS | BAS, FAS, EFAS |
| | History of AF | | BAS | BAS, FAS, EFAS |
| | Symptoms | | BAS | BAS, FAS, EFAS |
| | Concomitant Diseases | | BAS | BAS, FAS, EFAS |
| | Diagnostics | | BAS | BAS, FAS, EFAS |
| | Medications List | | BAS | BAS, FAS, EFAS |
| | AFEQT | | BAS | BAS, FAS, EFAS |
| | Anticoagulation (before/during first documented procedure) | ANCILLARY<br>OBJECTIVE | BAS | BAS, FAS, EFAS |
| FIRST<br>DOCUMENTED<br>PROCEDURE | Administrative information | | APS, BAS | APS, BAS, FAS,<br>EFAS |
| | Procedure summary information | ANCILLARY<br>OBJECTIVE | BAS | BAS, FAS, EFAS |
| | Consumables | | BAS | BAS, FAS, EFAS |
| | PVI confirmation | | BAS | BAS, FAS, EFAS |
| | Hospital discharge | | APS, BAS | APS, BAS, FAS,<br>EFAS |
| | Medication list at discharge | | BAS | BAS, FAS, EFAS |
| ADDITIONAL PROCEDURE(S) | Administrative information | | - | BAS, FAS, EFAS |
| | Procedure summary information | ANCILLARY<br>OBJECTIVE | - | BAS, FAS, EFAS |
| | Consumables | | - | BAS, FAS, EFAS |
| | PVI confirmation | | - | BAS, FAS, EFAS |
| STUDY EXIT | Study exit | | APS, BAS | APS, BAS, FAS,<br>EFAS |
| AE | Administrative Information/Adverse Event | ADDITIONAL OBJECTIVE | - | BAS, FAS, EFAS |
| | Relatedness of the AE | | - | BAS, FAS, EFAS |
| | Description of AE/AEAC | | - | BAS, FAS, EFAS |
| GENERAL FU | Administrative Information | | - | BAS, FAS, EFAS |
| | History of Arrhythmias since the last visit | | - | BAS, FAS, EFAS |

| | Diagnostics | | - | BAS, FAS, EFAS |
|---|---|---|---|---|
| | Symptoms | | - | BAS, FAS, EFAS |
| | Hospitalizations | | - | BAS, FAS, EFAS |
| | Medication List | | - | BAS, FAS, EFAS |
| 12MFU VISIT<br>12MFU B'<br>PHONE | / Administrative Information | | - | BAS, FAS, EFAS |
| | History of Arrhythmias since the last visit | MAIN<br>OBJECTIVE | - | BAS, FAS, EFAS |
| | Diagnostics | | - | BAS, FAS, EFAS |
| | Symptoms | | - | BAS, FAS, EFAS |
| | Hospitalizations | | - | BAS, FAS, EFAS |
| | Medication List | | - | BAS, FAS, EFAS |
| | AFEQT | ANCILLARY<br>OBJECTIVE | - | BAS, FAS, EFAS |

## **Appendix C: Subgroup analysis**

Predefined subgroups (V1.0)

| Subgroup description | Analysis set, additional inclusion or exclusion criteria | Tables and scope for analysis |
|---|---|---|
| Indication to schedule Phased RFA: Paroxysmal AF | FAS, EFAS incl.: excl.: | Baseline<br>First documented procedure<br>Additional procedure<br>12MFU |
| Indication to schedule Phased RFA: Persistent AF | FAS, EFAS | Baseline<br>First documented procedure<br>Additional procedure |
| reisistent Ai | incl.:<br>excl.: | 12MFU |
| Indication to schedule Phased RFA: Longstanding persistent AF | FAS, EFAS incl.: excl.: | Baseline<br>First documented procedure<br>Additional procedure<br>12MFU |
| Successful first documented procedure | FAS, EFAS incl.: excl.: | Baseline<br>First documented procedure<br>Additional procedure<br>12MFU |
| Non-successful first documented procedure | FAS, EFAS incl.: excl.: | Baseline<br>First documented procedure<br>Additional procedure<br>12MFU |
| First documented procedure: PVAC GOLD solely | FAS, EFAS incl.: Phased RFA catheters = PVAC GOLD, general number if catheters used = 1 excl.: adjunctive devices used during the procedure, disregarding sheaths used | First documented procedure<br>Additional procedure<br>GFU<br>12MFU |
| First documented procedure: PVAC GOLD + other catheters | FAS, EFAS incl.: Phased RFA catheters = PVAC GOLD, general number if catheters used > 1, additional Phased catheter used (MAAC, MASC and/or Other) excl.: adjunctive devices used during the procedure, disregarding sheaths used | First documented procedure<br>Additional procedure<br>GFU<br>12MFU |
| First documented procedure:<br>Phased RFA catheter solely | FAS, EFAS incl.: Phased RFA catheters used, general number if catheters used = 1 excl.: adjunctive devices used during the procedure, disregarding sheaths used | First documented procedure<br>Additional procedure<br>GFU<br>12MFU |
| First documented procedure: Phased RFA catheter + adjunctive devices | FAS, EFAS incl.: Phased RFA catheters = PVAC GOLD, general number if catheters used > 1, additional Phased catheter used (MAAC, MASC and/or Other), adjunctive devices used during the procedure excl.: | First documented procedure<br>Additional procedure<br>GFU<br>12MFU |
| Procedure: Patients with multiple procedures | FAS, EFAS | Baseline<br>First documented procedure<br>Additional procedure |

| | incl.: patients with > 1 documented procedure excl.: | GFU<br>12MFU |
|---|---|---|
| Baseline: Patient with AF surgery or ablations in history | FAS, EFAS incl.: prior AF surgery, status post ablation (endocardial, epicardial, Catheter PV, Phased RF, 3D RF or Other ablation technologies) excl.: | Baseline<br>First documented procedure<br>Additional procedure<br>GFU<br>12MFU |
| Baseline: Patient without AF surgery or ablations in history | FAS, EFAS incl.: no prior AF surgery, no status post ablation (endocardial, epicardial, Catheter PV, Phased RF, 3D RF or Other ablation technologies) excl.: | Baseline<br>First documented procedure<br>Additional procedure<br>GFU<br>12MFU |
| Baseline: Reveal implanted patients | FAS, EFAS incl.: ICM implantation - Reveal XT, Reveal LINQ or other excl.: | Baseline<br>First documented procedure<br>Additional procedure<br>GFU<br>12MFU |
| First documented procedure: Anticoagulation in patients with LAAO | FAS, EFAS incl.: LAAO implantation, anticoagulation medication prior first documented procedure excl.: | Baseline<br>First documented procedure<br>12MFU |
| First documented procedure: patients with LAAO | FAS, EFAS incl.: LAAO implantation excl.: anticoagulation medication prior first documented procedure | Baseline<br>First documented procedure<br>12MFU |
| Patients with administrated at least<br>one antiarrhythmic drug (except<br>beta-blocker) | FAS, EFAS incl.: patients with >=1 antiarrhythmic medication (except beta-blocker) at any time of this study excl.: | Baseline<br>First documented procedure<br>GFU<br>12MFU |
| Patients without antiarrhythmic drug therapy | FAS, EFAS incl.: no antiarrhythmic medication at any time of this study excl.: | Baseline<br>First documented procedure<br>GFU<br>12MFU |
| First documented procedure: Patients with discontinued oral anticoagulation before the procedure | FAS, EFAS incl.: patients with oral anticoagulation prior to scheduled phased RFA and discontinued before first documented procedure excl.: | First documented procedure<br>GFU<br>12MFU |
| First documented procedure: Patients with oral anticoagulation before the procedure | FAS, EFAS incl.: patients with oral anticoagulation prior to scheduled phased RFA and not discontinued before first documented procedure excl.: | First documented procedure<br>GFU<br>12MFU |
| Patients lost to 12 month FU | APS, BAS incl.: patients w/o 12MFU excl.: | Baseline<br>First documented procedure<br>Additional procedure<br>GFU<br>12MFU |

## **Appendix D: Analysis of comparison groups**

Predefined comparison groups (V1.0)

| Comparison description | Analysis set, additional inclusion or exclusion criteria | Tables and scope for analysis | At time of<br>Interim<br>analysis | At time<br>of Final<br>analysis |
|---|---|---|---|---|
| Age | FAS, EFAS | Baseline | - | X |
| <65, 65-74, ≥75 | incl.: Age available<br>excl.: | First documented procedure<br>Additional procedure<br>GFU<br>12MFU | | |
| Body Mass Index | FAS, EFAS | Baseline | - | Х |
| <18.5, 18.5 to <25, 25 to <30, ≥30 | incl.: BMI available<br>excl.: | First documented procedure<br>Additional procedure<br>GFU<br>12MFU | | |
| EHRA AF symptoms (at admission during the last 12 months) None, Yes – I "No", II "Mild", III "Severe", IV "Disabling" | FAS, EFAS incl.: AF symptoms available excl.: | Baseline<br>First documented procedure<br>Additional procedure<br>GFU<br>12MFU | - | X |
| <u> </u> | | | | |
| Gender<br>Males, Females | BAS, FAS, EFAS incl.: Gender available excl.: | Baseline<br>First documented procedure<br>Additional procedure<br>GFU<br>12MFU | × | X |
| First documented pro- | BAS, FAS, EFAS | First documented procedure | X | Х |
| Regular case, Training case | incl.: Regular or train-<br>ing case available<br>excl.: | Additional procedure<br>GFU<br>12MFU | | |
| Discharge after First<br>documented procedure<br>Patient discharged<br>home, Transferred to<br>another hospital, Death | FAS, EFAS incl.: Discharge available excl.: | First documented procedure<br>Additional procedure<br>GFU<br>12MFU | - | X |
| Adverse events | FAS, EFAS | First documented procedure | - | Х |
| Patients with AE during<br>12 months, Patients<br>w/o AE during 12<br>months | incl.: Adjudicated<br>events available<br>excl.: | Additional procedure<br>GFU<br>12MFU | | |
| Re-occurrence of AF | FAS, EFAS | Baseline<br>First documented procedure | - | Х |
| Patients with re-occur-<br>rence AF, Patients w/o<br>re-occurrence AF dur-<br>ing 12 months | incl.:<br>excl.: | GFU<br>12MFU | | |
| First documented pro- | BAS, FAS, EFAS | First documented procedure | X | Х |
| Phased RFA <40 min of<br>fluoroscopy time vs. >=<br>40 min of fluoroscopy<br>time | incl.: Fluoroscopy time<br>available<br>excl.: | Additional procedure<br>GFU<br>12MFU | | |
| First documented pro-<br>cedure | BAS, FAS, EFAS | First documented procedure<br>Additional procedure<br>GFU<br>12MFU | X | X |

| General time of the procedure time <100 min vs. >=100 min | incl.: Total procedure<br>time available<br>excl.: | | | |
|---|---|---|---|---|
| Patients with more than<br>5 GFU vs. all other pa-<br>tients | BAS, FAS, EFAS<br>incl.:<br>excl.: | Baseline<br>GFU<br>12MFU | - | Х |
| Patients lost to 12MFU<br>vs. not lost to 12MFU<br>(according SAP chap-<br>ter7) | BAS<br>incl.:<br>excl.: | Baseline<br>GFU<br>12MFU | - | X |
| Analysis of missed data | incl.:<br>excl.: | Full tables set | - | Х |
| DAP by country | incl.:<br>excl.: | Baseline | - | Х |
| Fluoroscopy time by country | BAS<br>incl.:<br>excl.: | Baseline | - | X |

## **Appendix E: Annotated eCRF V1.3 and V1.4**

## **Appendix F: Follow-up Re-Assignment**

| Issue | Decision | Center-Patient-ID |
|---|---|---|
| 12MFU outside 12MFU | Use GFU instead of 12MFU for analysis | 3580-1222, 4497-335, 4497-337, |
| time window and GFU | | 4497-345, 4497-1529, 9641-551 |
| inside | | |
| 12MFU outside 12M | Use 12MFU as GFU in 9-12M time win- | 1946-1671, 1946-1674, 1946-1678, |
| time window and no | dow analysis | 1946-1679, 2737-1642, 3140-463, |
| GFU inside | | 3580-1444, 4608-1472, 5042-820, |
| | | 5042-832, 5576-207, 5576-208, 5576- |
| | | 211, 5576-212, 5576-213, 5576-218, |
| | | 5576-219, 5576-1191, 5576-1193, |
| | | 7549-402, 7554-1319, 7626-859, |
| | | 7626-860, 7626-861, 7626-865, 7626- |
| Duplicate 12MFUs | Use 12MFU visit for 12M analysis and | 1579<br>8413-420 |
| (Visit and by Phone) in- | disregard 12MFU phone | 0413-420 |
| side 12M time window | disregard 121VII o priorie | |
| Side 12101 time window | | |
| 12MFU and GFU inside, | Use 12MFU for 12M analysis and dis- | 3580-1735, 3730-190, 3730-195, |
| events only in 12MFU | regard GFU | 4497-339, 4497-350, 4497-903, 4497- |
| and at most minor dif- | regard of o | 909, 4497-911, 4497-920, 4497-1107, |
| ferences | | 4497-1109, 4497-1119, 4497-1123, |
| | | 4497-1516, 4497-1714, 4497-1781, |
| | | 4497-1789, 4497-1801, 4497-1803, |
| | | 5658-175, 6021-633, 6807-86, 6979- |
| | | 497, 8533-147, 9641-1456, 9641- |
| | | 1457, 9641-1458, 9641-1461, 9641- |
| | | 1467 |
| 12MFU and GFU inside | Transfer event details (e.g. AF- | 3354-42, 3730-181, 4497-1102, 4497- |
| 12M time window, | reoccurrence, Hospitalisation) to | 1118, 9641-1463, 9641-1464, 9641- |
| events only in GFU and | 12MFU for analysis and disregard GFU | 2593 |
| at most minor differ- | | |
| ences | | |
| 12MFU and GFU inside | Use 12MFU for analysis and transfer | 4497-1126, 4497-1523, 5658-164, |
| 12M time window, dif- | events from GFU | 6979-585, 9641-1455, 9641-2601 |
| ferent events and mi- | | |
| nor differences in | | |
| 12MFU and GFU | | |

#### This Statistical Analysis Plan has been written with reference to:

ICH GCP E6: International Conference on Harmonisation Guideline for Good Clinical Practice

ICH GCP E9: International Conference on Harmonisation Statistical Principles for Clinical Trials

Directive 2001/20/EC

MPG Medizinproduktegesetz

MPKV Verordnung über klinische Prüfungen von Medizinprodukten